CLINICAL TRIAL: NCT03931083
Title: Screening Test Accuracy of a Gynocular™, HR-HPV Testing, and VIA for Detection of Cervical Intraepithelial Neoplasia, Grade Two and Above, in Women Living With HIV in Lusaka, Zambia
Brief Title: Screening Test Accuracy of Gynocular™, HR-HPV Testing, VIA for Detection of Cervical Neoplastic Lesions, in Women Living With HIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bern (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other); Cervical Cancer Prevention Program in Zambia (Unknown); International Agency for Research on Cancer (Other)
Responsible Party: Sponsor
Other Study IDs: GYNOCULAR; KFS-4156-02-2017 (Other Grant/Funding Number: Swiss Cancer Research); Esther17G9 (Other Grant/Funding Number: ESTHER Switzerland); U01AI069924 (NIH)
Record Dates: First submitted 2019-04-15; First posted 2019-04-30 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Uterine Cervical Neoplasms; HIV/AIDS
MeSH Terms: conditions — Uterine Cervical Neoplasms; Acquired Immunodeficiency Syndrome | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For a biopsy, a very small sample (appr. 2X2X1 mm3) of tissue is taken from the cervix. The study nurse will take the biopsies after the Gynocular™ exam. Biopsies are taken of all acetowhite lesions. If no lesions are seen, a total of 4 biopsies will be taken within the transformation zone (12, 3, 6 and 9 o' clock positions). Bleeding is minimal, the biopsy site does not require stitches. The length of time it takes for this to heal varies but can be approximately 7 days. If the study participant informs the study nurse of any biopsy-related adverse event (AE), the study nurse will record this information in the study-specific data collection tool for AEs. The clinical team will manage the AE according to national guidelines and follow-up with the participant until the event is resolved.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Portable magnification device (Gynocular™): The Gynocular™ examination will be performed following the steps involved in colposcopy as described in the IARC colposcopy manual. These steps include: visualization of the vagina, vulva and cervix following insertion of a speculum, magnified assessment after application of normal saline, examination of cervical vessel patterns using the red-free mode (or green filter), application of 5% acetic acid for 1 minute and finally assessment following application with Lugol's iodine. The findings of the live examination will be documented using the parameters of the Swede score. Each parameter is scored between zero and two. Treatment will be based on the results found at histopathology, unless the woman is also VIA positive in which case, after biopsy she will undergo routine treatment as per local guidelines. The results will be used to determine the optimal threshold for treatment in WLHIV.
  Interventions: Diagnostic Test: Screening for CIN2+/HSIL
- Testing for high risk HPV (HRHPV): To reduce the number of examinations undergone by the study participant during the same day, HRHPV testing will be carried out at the time of the first gynecological examination by the VIA nurse (see next arm). Using specific single-use cervical cytobrush provided by GeneXpert, a specimen will be collected immediately prior to VIA examination. Cervical cytobrush specimens will be placed into ThinPrep PreservCyt (Cepheid, Sunnyvale, CA) immediately after collection. The HR-HPV testing of cervical specimens will be conducted by a GeneXpert™ machine (Cepheid, Sunnyvale, CA), which will be placed at the health facility and will be operated by a trained nurse in accordance with the manufacturer's instructions. Additionally, as part of the baseline clinical characteristics of the study participant, the study participant will undergo an STI test at the same time. The sample will be collected and tested using the same GeneXpertTM platform.
  Interventions: Diagnostic Test: Screening for CIN2+/HSIL
- Visual inspection with acetic acid (VIA): VIA, which is standard of care for cervical cancer screening in Zambia, will be carried out using the methodology described by IARC. This is summarized as follows: visualization of the vagina, vulva and cervix following insertion of a speculum; assessment with the naked eye after application of normal saline; and further assessment after application of 5% acetic acid for 1 minute. This will be recorded as normal or abnormal by the assessor.
  Interventions: Diagnostic Test: Screening for CIN2+/HSIL
- Histopathological examination of tissue biopsies: All acetowhite lesions will be biopsied. When no lesion is seen, one biopsy is taken from each quadrant at the squamocolumnar junction. Biopsies will be sent and examined in a South African based lab. All histological slides will also be verified independently by an IARC trained pathologist at the end of the study. Histological endpoints are defined by the CIN classification system: CIN 1 affects only the lower third of the epithelium (mild dysplasia), CIN 2 involves two thirds of the epithelium and CIN 3 involves the full thickness (severe dysplasia and carcinoma in situ). These findings can be dichotomized by the Lower Anogenital Squamous Terminology into low-grade squamous intraepithelial lesions (LSIL) and high-grade squamous intraepithelial lesions (HSIL). All patients with CIN grade 2 that stained diffusely positive for p16 are considered as HSIL, all patients with CIN 3 are considered as HSIL. Expression of p16 will be visually assessed by immunohistochemistry.
  Interventions: Diagnostic Test: Screening for CIN2+/HSIL

INTERVENTIONS:
Diagnostic Test: Screening for CIN2+/HSIL — The investigators will compare three different screening methods: visual assessment with portable magnification device , visual inspection after application of acetic acid, screening for high risk variants of HPV. All patients will receive cervical biopsies and histopathological examination.

SUMMARY:
Cervical cancer in HIV-positive women is largely preventable through regular screening. The World Health Organization (WHO) recommends cervical screening for HIV-positive women every three years. Currently the least costly method for screening and the most viable option for many countries is visual inspection after application of acetic acid (VIA). Alternative testing methods are HPV testing and assessment with a portable magnification device. The investigators plan to assess and compare the screening test accuracy of these screening tests in women living with HIV. All women will receive histopathology reference standard.

DETAILED DESCRIPTION:
The simplest and least costly method for cervical cancer screening is visual inspection after application of acetic acid (VIA). However, the ability of this screening method to correctly identify precancerous lesions (sensitivity) and women free from these lesions (specificity) is limited. The investigators aim to identify alternative screening methods which maximize sensitivity and specificity, particularly in HIV-infected women in receiving care in Southern Africa. The investigators will evaluate the screening test accuracy of a new portable magnification device , the Gynocular™ with Swede score assessment, in women who are HIV-positive and eligible for cervical cancer screening. The investigators will assess the accuracy of the device when used as a stand alone test, as well as when used subsequent to positive VIA or HPV tests. The investigators will make comparisons with current screening practices (VIA alone), as well as, recommended screening practices (HPV testing). The investigators will enrol 450 HIV-positive women receiving care for HIV/AIDS at the Centre for Infectious Disease Research in Zambia, in Lusaka, Zambia. Consenting women will be screened with VIA, HPV testing and visual assessment with Gynocular™. All women undergo biopsy (reference standard) and receive treatment as indicated and in accordance with national guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected women confirmed through medical records
2. Women residing within Lusaka district and plans to stay in this area for the next 6 months
3. Women between 18 and 65 years of age (age bracket as per Zambian guidelines for cervical cancer screening)
4. Able and willing to consent
5. Willing to undergo a pelvic examination and cancer screening
6. Has had sexual intercourse before
7. Agrees to have follow-up appointment in 6 months

Exclusion Criteria:

1. Women with a history of cervical cancer or previous hysterectomy (where the cervix was also removed)
2. Pregnant women or women who plan to get pregnant within the next 6 months
3. Women who have been vaccinated against HR-HPV

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Study Population: The study population includes women who are enrolled in the ART program at Kanyama Clinic, Lusaka, Zambia. Kanyama Clinic is situated on the western side of the central business district, 3km away from the town centre. It has a catchment population of 262,715. It has registered 52,658 people living with HIV, of which 40,650 have commenced treatment. In addition to ART services, the clinic has also been providing cervical cancer screening since October 2006. The clinic is well established in the application of cancer screening based on a "screen-and-treat" approach, where women undergo visual screening, followed by immediate treatment where possible. Since inception in 2006, the clinic has screened over 23,900 women for cervical cancer. Clinic nurses are trained to offer cervical cancer screening and treatment with cryotherapy or thermal coagulation and to refer suspicious cases for LEEP and further treatment.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Test accuracy (sensitivity, specificity) of the Gynocular™ when used as stand-alone tests to detect CIN2+ | 6 months
  To estimate the sensitivity and specificity of the Gynocular when used as a standalone tests to detect CIN2+ among WLHIV.
Test accuracy (sensitivity, specificity) of HR-HPV when used as stand-alone tests to detect CIN2+ | 6 months
  To estimate the sensitivity and specificity of HR-HPV when used as a standalone tests to detect CIN2+ among WLHIV.
Test accuracy (sensitivity, specificity) of VIA when used as stand-alone tests to detect CIN2+ | 6 months
  To estimate the sensitivity and specificity of VIA when used as a standalone tests to detect CIN2+ among WLHIV.

SECONDARY OUTCOMES:
Diagnostic test accuracy of the Gynocular™to detect CIN2+/HSIL: other estimates, stand alone | 6 months
  To determine other estimates of test accuracy of the Gynocular™ (including positive and negative predictive values, positive and negative likelihood ratios, false positive rate, false negative rate, number needed to screen and area under the ROC curve (AUC).
Diagnostic test accuracy of HR-HPV testing to detect CIN2+/HSIL: other estimates, stand alone | 6 months
  To determine other estimates of HR-HPV testing test accuracy (including positive and negative predictive values, positive and negative likelihood ratios, false positive rate, false negative rate, number needed to screen and area under the ROC curve (AUC).
Diagnostic test accuracy of VIA to detect CIN2+/HSIL: other estimates, stand alone | 6 months
  To determine other estimates of VIA test accuracy (including positive and negative predictive values, positive and negative likelihood ratios, false positive rate, false negative rate, number needed to screen and area under the ROC curve (AUC).
Diagnostic test accuracy of HR-HPV testing followed by Gynocular™ to detect CIN2+/HSIL: test combination | 6 months
  To determine estimates of test accuracy for combinations of screening tests, i.e. HR-HPV followed by Gynocular™
Diagnostic test accuracy of HR-HPV testing followed by Gynocular™ to detect CIN2+/HSIL: test combination - subgroup analyses | 6 months
  To investigate the effects of age, menopause, parity, ART status, HIV RNA, education, contraception, CD4 cell count, previous treatment for precancerous disease and sexually transmitted infections (STIs) on test accuracy of test combination in subgroup analyses
Diagnostic test accuracy of the Gynocular™ followed by HR-HPV testing to detect CIN2+/HSIL: test combination | 6 months
  To determine estimates of test accuracy for combinations of screening tests, i.e. Gynocular™ followed by HR-HPV
Diagnostic test accuracy of the Gynocular™ followed by HR-HPV testing to detect CIN2+/HSIL: test combination subgroup analyses | 6 months
  To investigate the effects of age, menopause, parity, ART status, HIV RNA, education, contraception, CD4 cell count, previous treatment for precancerous disease and sexually transmitted infections (STIs) on test accuracy of test combination in subgroup analyses
Diagnostic test accuracy VIA followed by Gynocular™ to detect CIN2+/HSIL: test combination | 6 months
  To determine estimates of test accuracy for combinations of screening tests, i.e. VIA followed by Gynocular™
Diagnostic test accuracy VIA followed by Gynocular™ to detect CIN2+/HSIL: test combination - subgroup analyses | 6 months
  To investigate the effects of age, menopause, parity, ART status, HIV RNA, education, contraception, CD4 cell count, previous treatment for precancerous disease and sexually transmitted infections (STIs) on test accuracy of test combination in subgroup analyses
Diagnostic test accuracy of the Gynocular™ followed by VIA to detect CIN2+/HSIL: test combination | 6 months
  To determine estimates of test accuracy for combinations of screening tests, i.e. Gynocular™ followed by VIA
Diagnostic test accuracy of the Gynocular™ followed by VIA to detect CIN2+/HSIL: test combination - subgroup analyses | 6 months
  To investigate the effects of age, menopause, parity, ART status, HIV RNA, education, contraception, CD4 cell count, previous treatment for precancerous disease and sexually transmitted infections (STIs) on test accuracy of test combination in subgroup analyses
Diagnostic test accuracy of the HR-HPV followed by VIA to detect CIN2+/HSIL: test combination | 6 months
  To determine estimates of test accuracy for combinations of screening tests: HR-HPV followed by VIA.
Diagnostic test accuracy of the HR-HPV followed by VIA to detect CIN2+/HSIL: test combination - subgroup analyses | 6 months
  To investigate the effects of age, menopause, parity, ART status, HIV RNA, education, contraception, CD4 cell count, previous treatment for precancerous disease and sexually transmitted infections (STIs) on test accuracy of test combination in subgroup analyses
Diagnostic test accuracy of the VIA followed by HR-HPV to detect CIN2+/HSIL: test combination | 6 months
  To determine estimates of test accuracy for combinations of screening tests: VIA followed by HR-HPV.
Diagnostic test accuracy of the VIA followed by HR-HPV to detect CIN2+/HSIL: test combination subgroup analyses | 6 months
  To investigate the effects of age, menopause, parity, ART status, HIV RNA, education, contraception, CD4 cell count, previous treatment for precancerous disease and sexually transmitted infections (STIs) on test accuracy of test combination in subgroup analyses
Subgroup analyses for the diagnostic test accuracy of Gynocular™: stand alone test | 6 months
  To investigate the effects of a age, menopause, parity, ART status, HIV RNA, education, contraception, CD4 cell count, previous treatment for precancerous disease and sexually transmitted infections (STIs) on test accuracy of test combination in subgroup analyses.
Subgroup analyses for the diagnostic test accuracy of VIA: stand alone test | 6 months
  To investigate the effects of age, menopause, parity, ART status, HIV RNA, education, contraception, CD4 cell count, previous treatment for precancerous disease and sexually transmitted infections (STIs) on test accuracy of test combination in subgroup analyses.
Subgroup analyses for the diagnostic test accuracy of HR-HPV testing: stand alone test | 6 months
  To investigate the effects of age, menopause, parity, ART status, HIV RNA, education, contraception, CD4 cell count, previous treatment for precancerous disease and sexually transmitted infections (STIs) on test accuracy of test combination in subgroup analyses
Subgroup analyses for the diagnostic test accuracy of VIA, HR-HPV testing and Gynocular™: Combined tests | 6 months
  To investigate the effects of age, menopause, parity, ART status, HIV RNA, education, contraception, CD4 cell count, previous treatment for precancerous disease and sexually transmitted infections (STIs) on test accuracy of test combination in subgroup analyses
Investigation of Swede Score in WLHIV | 6 months
  Area under the receiver operating characteristic (ROC) curve for Swede score determined by Gynocular™ in WLHIV
Investigation of co-infections of premalignant and malignant disease (STIs/HR-HPV) | 6 months
  Descriptive analysis of the STI and HR-HPV type distribution associated with each stage of CIN, and when there is persistent disease in WLHIV.
Investigation of Trichomonas vaginalis prevalence and persistence in association with menstrual hygiene practices | 6 months
  Descriptive analysis of the prevalence and persistence of Trichomonas vaginalis in association with vaginal and menstrual hygiene practices.
Investigations to inform telemedicine capacity: Comparison of image quality | 6 months
  Description of image quality from static assessors, in terms of the assessors' ability to adequately evaluate the images.
Investigations to inform telemedicine capacity: use of static images | 6 months
  Proportion of correctly diagnosed CIN2+ through static images obtained by the Gynocular™.
Investigations to inform telemedicine capacity: ROC curve for Swede score | 6 months
  Area under the ROC for static image Swede score obtained by Gynocular™ in WLHIV.
Investigations to inform telemedicine capacity: Live versus static assessors | 6 months
  Cohen's kappa coefficient to assess agreement between live and static assessors.
Artificial Intelligence (AI) for improving the detection of precancerous cervical lesions: testing AI algorithm | 6 months
  Test accuracies of AI deep learning tool retrospectively using coded images obtained in the study through the Gynocular™ and smartphone.
Artificial Intelligence for improving the detection of precancerous cervical lesions: improve AI algorithm | 6 months
  Inform and improve AI deep learning tools to detect HSIL by using images or GIFs obtained in the study through the Gynocular™ and smartphone.
Diagnostic test accuracy of AI tool to detect CIN2+/HSIL: other estimates, stand alone | 6 months
  To estimate the sensitivity and specificity of HR-HPV when used as a standalone tests to detect CIN2+/HSIL among WLHIV.
Diagnostic test accuracy of HR-HPV testing followed by AI tool to detect CIN2+/HSIL: test combination | 6 months
  To determine estimates of test accuracy for combinations of screening tests, i.e. HR-HPV followed by AI tool

OTHER OUTCOMES:
Safety outcomes: For each adverse event found the investigators will calculate crude frequencies | 9 months
  Adverse events will be recorded. The investigators will ask participants to inform the study nurse or assistant if they develop any of these, in person or by phone. Given the health system in this context is not centralized, it is most efficient to ask participants to report these to the clinical team and investigators. Information describing these events will include: time of onset, duration, resolution, action to be taken, assessment of intensity, relationship with study treatment. The clinical team will also complete assessments of seriousness, causality and expectedness. Participants are asked to inform the clinical team immediately if any AE occur in the 9 months following their initial enrolment. At each visit, the Study nurse/assistant will also inquire about any adverse events that have occurred, for verification. For each adverse event found the investigators will calculate crude frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Bohlius, MD, Principal Investigator — julia.bohlius@ispm.unibe.ch
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided
We plan to publish results in open access journals with data available in accordance with FAIR principles.

REFERENCES:
- [Derived] Taghavi K, Moono M, Mwanahamuntu M, Roumet M, Limacher A, Kapesa H, Madliwa T, Rutjes A, Basu P, Low N, Manasyan A, Bohlius J. Accuracy of screening tests for cervical precancer in women living with HIV in low-resource settings: a paired prospective study in Lusaka, Zambia. BMJ Oncol. 2024 Feb 10;3(1):e000111. doi: 10.1136/bmjonc-2023-000111. eCollection 2024. PMID 39886160
- [Derived] Taghavi K, Moono M, Mwanahamuntu M, Roumet M, Limacher A, Kapesa H, Madliwa T, Rutjes A, Basu P, Low N, Manasyan A, Bohlius J. Accuracy of screening tests for cervical pre-cancer in women living with HIV in low-resource settings: a paired prospective study in Lusaka, Zambia. medRxiv [Preprint]. 2023 Jun 1:2023.05.31.23290779. doi: 10.1101/2023.05.31.23290779. PMID 37398043
- [Derived] Taghavi K, Moono M, Mwanahamuntu M, Basu P, Limacher A, Tembo T, Kapesa H, Hamusonde K, Asangbeh S, Sznitman R, Low N, Manasyan A, Bohlius J. Screening test accuracy to improve detection of precancerous lesions of the cervix in women living with HIV: a study protocol. BMJ Open. 2020 Dec 18;10(12):e037955. doi: 10.1136/bmjopen-2020-037955. PMID 33371015

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT03931083/SAP_000.pdf